CLINICAL TRIAL: NCT04489758
Title: Utility of a Novel Imaging Algorithm (4DX) for the Diagnosis of Constrictive Bronchiolitis
Brief Title: 4DX for the Diagnosis of Constrictive Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: 4DMedical (Industry)
Responsible Party: Principal Investigator, Bradley Richmond, Assistant Professor of Pulmonary/Critical Care Medicine, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 200473
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Constrictive Bronchiolitis
Keywords: fluoroscopy; X-ray velocimetry
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Intervention Model Description: 4Dx XV Ventilation Analysis applied to fluoroscopic images
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constrictive Bronchiolitis (Experimental): Veterans with surgical lung biopsy-proven constrictive bronchiolitis
  Interventions: Diagnostic Test: X-ray velocimetry analyzed by 4Dx XV Ventilation Analysis
- Controls (Active Comparator): Control patients with minimal smoking history and no chronic lung disease or respiratory symptoms
  Interventions: Diagnostic Test: X-ray velocimetry analyzed by 4Dx XV Ventilation Analysis

INTERVENTIONS:
Diagnostic Test: X-ray velocimetry analyzed by 4Dx XV Ventilation Analysis — Fluoroscopy will be performed for a complete tidal breath and full exhalation at 5 angles (AP, +/- 36 degrees from AP, and +/- 72 degrees from AP) while the patient's arms are raised overhead. 4Dx XV Ventilation Analysis software will be used to analyze these images. Both groups will also undergo pulmonary function testing and take a questionnaire regarding respiratory symptoms.

SUMMARY:
Constrictive bronchiolitis is an uncommon lung disease that has been described in Veterans of conflicts in Iraq and Afghanistan. Although these Veterans have evidence of constrictive bronchiolitis on lung biopsies, non-invasive tests such as pulmonary function tests (PFTs) are often normal. This study will determine whether analysis of fluoroscopy images using the 4Dx XV Ventilation Analysis software developed by 4D Medical will be able to detect constrictive bronchiolitis in Veterans better than PFTs.

DETAILED DESCRIPTION:
Constrictive (or obliterative) bronchiolitis is a rare pulmonary disease characterized by subepithelial inflammatory and fibrotic narrowing of the bronchioles on histologic analysis, which often presents with nonspecific symptoms such as progressive dyspnea on exertion and nonproductive cough over weeks to months. Constrictive bronchiolitis may be triggered by autoimmune disease, chronic allograft rejection in lung transplant recipients, graft versus host disease in stem cell transplant recipients, viral illness, or inhaled toxins. Although pulmonary function tests (PFTs) may be helpful for the diagnosis of constrictive bronchiolitis, a study performed by King and colleagues in 2009 found that many Veterans with biopsy-proven constrictive bronchiolitis had normal PFTs. Thus, for these patients, more sensitive methods of noninvasive testing are needed.

4Dx XV Ventilation Analysis is a new imaging analysis algorithm which utilizes standard fluoroscopy to quantify ventilation with sufficient fidelity to identify regional differences. Fluoroscopic images of a single tidal breath are obtained at 5 distinct angles (direct AP, +/- 36 degrees, and +/- 72 degrees). Readouts from the 4Dx XV Ventilation Analysis include absolute value of total lung ventilation, heterogeneity of lung ventilation, a frequency distribution of lung ventilation as a line plot, and a regional map of lung ventilation. In addition, an expiratory time constant (time to exhale 63% of the tidal volume), heterogeneity of the expiratory time constant, frequency distribution of expiratory time constant as a line plot, and a regional map of expiratory time constant are also calculated. Pilot studies performed by 4D Medical show data generated by the 4Dx XV Ventilation Analysis software applied to fluoroscopy is reproducible in individuals with normal lung function and the heterogeneity index increases in individuals undergoing radiation therapy.

The investigators hypothesize that the 4Dx XV Ventilation Analysis program, when applied to standard fluoroscopic images, is more sensitive for the diagnosis of constrictive bronchiolitis than PFTs in Veterans with constrictive bronchiolitis. Specific metrics that will be evaluated with the software include ventilation heterogeneity and expiratory phase constants, among other metrics. Endpoints will be compared during tidal breathing and a full exhalation to residual volume from functional residual capacity.

ELIGIBILITY:
Inclusion Criteria

Constrictive bronchiolitis arm:

* Biopsy demonstrating constrictive bronchiolitis
* Prior CT Chest
* 18-60 years old
* < 1 pack year history of tobacco use

Control arm:

* 18-60 years old
* Prior CT Chest without evidence chronic lung disease as judged by a Pulmonologist
* No clinically significant dyspnea or functional limitations
* < 1 pack year history of tobacco use

Exclusion Criteria (for both arms)

* Pregnancy (as determined by testing on the morning prior to fluoroscopy)
* Inability to undergo PFTs or fluoroscopy
* Inability to raise arms above a 90-degree angle

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
X-ray velocimetry results | 1 month
  Heterogeneity of ventilation as detected by X-ray velocimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King MS, Eisenberg R, Newman JH, Tolle JJ, Harrell FE Jr, Nian H, Ninan M, Lambright ES, Sheller JR, Johnson JE, Miller RF. Constrictive bronchiolitis in soldiers returning from Iraq and Afghanistan. N Engl J Med. 2011 Jul 21;365(3):222-30. doi: 10.1056/NEJMoa1101388. PMID 21774710
- [Derived] Richmond BW, Lester MG, Lui V, Dusting J, Raju S, Snell GI, Blackburn JB, Douglas K, Miller RF, Siddharthan T, Fouras A. X-ray velocimetry provides temporally and spatially-resolved biomarkers of lung ventilation in small airways disease. Respir Res. 2025 Jul 2;26(1):226. doi: 10.1186/s12931-025-03295-6. PMID 40604808